CLINICAL TRIAL: NCT07232446
Title: Effect of Vulvar Re-Antisepsis Before Cystoscopy on Urinary Infections in Laparoscopic Hysterectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Alaattin Karabulut (Other)
Responsible Party: Sponsor-Investigator, Alaattin Karabulut, Principal Investigator, Tepecik Training and Research Hospital
Organization: Tepecik Training and Research Hospital (Other)
Other Study IDs: TepecikTRH-AKarabulut-002
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Urinary Tract Infection; Laparoscopic Hysterectomy; Cystoscopy; Antisepsis
Keywords: vulvar antisepsis; cystoscopy; Laparoscopic Hysterectomy; Urinary Tract Infection; Infection Prevention
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Antisepsis: Patients undergoing total laparoscopic hysterectomy who receive routine preoperative vulvar antisepsis only. Cystoscopy is performed at the end of the procedure using carbon dioxide (CO₂) as the distension medium, without any additional re-antisepsis before cystoscope insertion.
- Re-Antisepsis Before Cystoscopy: Patients undergoing total laparoscopic hysterectomy who receive additional vulvar re-antisepsis immediately before intraoperative cystoscopy. The cystoscopy is performed using carbon dioxide (CO₂) as the distension medium to evaluate bladder integrity and ureteral jets.
  Interventions: Procedure: Additional Vulvar Re-Antisepsis Before Cystoscopy

INTERVENTIONS:
Procedure: Additional Vulvar Re-Antisepsis Before Cystoscopy — In this observational cohort, some patients receive an additional vulvar re-antisepsis immediately before intraoperative cystoscopy during total laparoscopic hysterectomy. The antisepsis is performed using standard povidone-iodine solution prior to cystoscope insertion. Cystoscopy is conducted using carbon dioxide (CO₂) as the distension medium.
  Groups: Re-Antisepsis Before Cystoscopy

SUMMARY:
This prospective observational study aims to evaluate whether additional vulvar re-antisepsis before intraoperative cystoscopy reduces the incidence of postoperative urinary tract infections (UTIs) in patients undergoing total laparoscopic hysterectomy for benign indications. In our institution, cystoscopy is routinely performed at the end of laparoscopic hysterectomy using carbon dioxide (CO₂) as the distension medium to assess bladder integrity and ureteral jet flow. However, potential contamination from the vaginal flora during cystoscopy may increase the risk of postoperative UTI. The study will compare two groups of patients: those receiving standard preoperative antisepsis only and those undergoing additional vulvar re-antisepsis immediately before cystoscopy. The primary outcome is the incidence of postoperative UTI diagnosed according to CDC criteria. Secondary outcomes include cystoscopy duration, catheterization time, and need for postoperative antibiotic therapy. Findings from this study may help determine whether an additional antisepsis step can improve infection control during laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is one of the most common postoperative complications following gynecologic surgery. In our institution, intraoperative cystoscopy is routinely performed during total laparoscopic hysterectomy (TLH) to assess bladder and ureteral integrity and to enable early detection of possible injuries. In our clinic, cystoscopy is performed using carbon dioxide (CO₂) as the distension medium. However, contamination of the cystoscope or instruments with vaginal flora during insertion may contribute to postoperative infections.

This prospective observational study aims to investigate whether performing additional vulvar re-antisepsis immediately before cystoscopy reduces postoperative UTI rates in patients undergoing TLH for benign indications.

Participants will be adult women undergoing TLH with intraoperative cystoscopy. The study population will be divided into two groups:

Group 1: Standard preoperative antisepsis only Group 2: Additional vulvar re-antisepsis performed immediately before cystoscopy

The primary outcome measure will be the incidence of postoperative UTI diagnosed in the early postoperative period according to CDC/NHSN criteria. Secondary outcomes will include cystoscopy duration, duration of urinary catheterization, and the need for postoperative antibiotic therapy.

All data will be collected prospectively using standardized case report forms. The findings of this study are expected to clarify whether a simple additional antisepsis step can effectively reduce postoperative UTIs without increasing operative time or procedural complexity, thereby contributing to infection control strategies during laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older
* Undergoing total laparoscopic hysterectomy (TLH) for benign gynecologic indications
* Intraoperative cystoscopy planned as part of the surgical procedure
* No evidence of urinary tract infection before surgery
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Positive preoperative urine culture
* Known immunodeficiency or current use of immunosuppressive therapy
* Patients with diabetes mellitus whose blood glucose levels are poorly controlled
* History of bladder or ureteral anatomical anomalies
* Cases converted to another surgical route or completed via the vaginal route
* Patients whose final pathology reveals malignant disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: dult women (≥18 years) undergoing total laparoscopic hysterectomy for benign gynecologic indications at the University of Health Sciences Tepecik Training and Research Hospital Department of Gynecology and Obsterics.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Urinary Tract Infection (CDC/NHSN Criteria) | Within 6 weeks after surgery
  Proportion of participants who develop a postoperative urinary tract infection (UTI) within 6 weeks after total laparoscopic hysterectomy, defined according to CDC/NHSN criteria (symptoms and signs consistent with UTI plus laboratory confirmation on urine testing or culture). Asymptomatic bacteriuria will not be counted as UTI. Diagnosis will be based on clinical follow-up evaluations, electronic medical records, and microbiology reports.

SECONDARY OUTCOMES:
Total Time Required for Cystoscopy Procedure Including Re-Antisepsis Step | From the start of cystoscopy preparation to removal of the cystoscope (typically 2-5 minutes).
  During surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Tepecik Training and Research Hospital, Department of Obstetrics and Gynecology, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared publicly. Summary-level data may be available upon reasonable request after publication of the study results.